CLINICAL TRIAL: NCT04196465
Title: Phase II Study of Neoadjuvant Immune Checkpoint Inhibitor in Patients With Resectable Gastrointestinal Cancers(Neo-Chance Study)
Brief Title: Phase II Study of Neoadjuvant Immune Checkpoint Inhibitor in Patients With Resectable Gastrointestinal Cancers
Acronym: NeoChance
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Sook Ryun Park, Associated professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0988
Record Dates: First submitted 2019-08-28; First posted 2019-12-12 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Subjects With Resectable and Localized Gastric Cancer; Subjects With Resectable Esophageal Cancer or Liver Cancer; Subjects With Resectable Liver Cancer
MeSH Terms: conditions — Liver Neoplasms | interventions — IMC-001

STUDY DESIGN:
Intervention Model Description: This study is a prospective, IMC-001 single arm, open label, single center, phase II study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Neoadjuvant IMC-001 (Experimental): Neoadjuvant immune check point inhibitor of IMC-001 in participants with resectable and localized gastric cancer, esophageal cancer, and hepatocellular carcinoma
  Interventions: Drug: IMC-001

INTERVENTIONS:
Drug: IMC-001 — IMC-001 is a fully human anti-programmed cell death ligand 1 (PD-L1) recombinant monoclonal antibody that strongly binds to PD-L1 to inhibit its binding to programmed cell death protein 1 (PD-1) or B7-1 (CD80). IMC-001 showed robust dose-dependent efficacy in animal models and no evidence of toxicity in cynomolgus monkeys

SUMMARY:
This is a phase II, open-label, prospective single-centered study. Subjects who meet the inclusion/exclusion criteria will be allocated to appropriate cohorts: 1) gastric cancer, 2) esophageal cancer and 3) hepatocellular carcinoma. Each cancer cohort group will be treated with two cycles of neoadjuvant immune checkpoint inhibitor of IMC-001 (1 cycle = 2 weeks) followed by curative resection and be followed up consecutively.

DETAILED DESCRIPTION:
This is a phase II, open-label, prospective single-centered study. Subjects who meet the inclusion/exclusion criteria will be allocated to appropriate cohorts: 1) gastric cancer, 2) esophageal cancer and 3) hepatocellular carcinoma. Each cancer cohort group will be treated with two cycles of neoadjuvant immune checkpoint inhibitor of IMC-001 (1 cycle = 2 weeks) followed by curative resection and be followed up consecutively.

The sample size of the study is determined based on a major pathologic response rate (primary endpoint) and by using Simon's single stage design from the subjects who receive preoperative neoadjuvant therapy of IMC-001.

In each cancer cohort group, the null and alternative response rates are assumed as 5% and 20%, respectively. This provides a power of 80% when calculating the difference between major pathologic response rates of 5% and 20% in two-tailed significance level of 0.153 (Type I error[two-tailed] of 15.3%). In order to reject the null hypothesis, at least two major pathological respondents are needed among 14 assessable subjects for each cancer cohort. After choosing the margin of safety as 10%, each cancer cohort will require 16 subjects and therefore a total of 48 subjects will be enrolled into the study.

ELIGIBILITY:
Inclusion Criteria:

<Disease-related inclusion criteria>

1. Histologically confirmed localized gastric adenocarcinoma, esophageal squamous cell carcinoma, hepatocellular carcinoma or clinically diagnosed hepatocellular carcinoma according to American Association for the Study of Liver Disease (AASLD) guidelines.However, in cases of hepatic carcinoma that can be clinically diagnosed according to AASLD guideline, no biopsy is performed.
2. Curatively resectable gastric adenocarcinoma, esophageal squamous cell carcinoma or hepatocellular carcinoma

   A. Gastric adenocarcinoma: clinical stage ≥T2 or regional lymph node metastasis (N+) (AJCC 8th)

   B. Esophageal squamous cell carcinoma: clinical stage ≥T1b or N+ (AJCC 8th)

   C. Hepatocellular carcinoma: a single hepatocellular carcinoma limited to liver or 3 or less hepatocellular carcinoma limited to liver without invasion to main portal trunk
3. The requirements for hematology, blood chemistry, and functionality in major organs are as follows (should be met within 7 days prior to the first administration of investigational medicinal product):

   A. Absolute neutrophil count ≥1,000/μL

   B. Platelets count ≥75,000/μL

   C. Total bilirubin ≤1.5 × Upper limit of Normal (ULN) (subjects with Gilbert syndrome: bilirubin ≤ 3.0 × ULN)

   D. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤ 2.5 × ULN; alkaline phosphatase ≤ 2.5 × ULN

   E. Serum creatinine ≤1.5 × ULN or creatinine clearance ≥50 mL/minute (creatinine clearance is first calculated by the formula of Cockcroft-Gault and in case of the value less than 50 mL/min, by collecting and examining 24-hour urine the subjects with the creatine clearance ≥50 mL/minute can be enrolled) (Refer to Supplement 1).

   F. Urine protein-creatinine ratio (UPC) ≤1 (in case of UPC >1, by collecting and examining 24-hour urine the subjects with the urine protein <2 g/day can be enrolled)

   G. Also, in case of hepatocellular carcinoma, liver function with Child-Pugh grade A (Refer to Supplement 2) and encephalopathy grade 0.
4. Measurable or evaluable lesion(s) according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (Refer to Supplement 3).
5. Tumor tissue specimen, classified as appropriate for biomarker analysis, must be provided (in case of hepatocellular carcinoma, subjects, without tissue specimen prior to the administration of investigational medicinal product, are allowed for enrollment into the study).

   <General inclusion criteria>
6. Aged ≥ 19 years old
7. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
8. Signed informed consent form
9. In the case of fertility men and women, Those who should be using adequate contraceptive measures while on study drug and for 3months following the last dose of study drug.

Exclusion Criteria:

<Tumor-related exclusion criteria>

1. Curatively unresectable or metastatic disease
2. Any prior treatment for gastric adenocarcinoma, esophageal squamous cell carcinoma or hepatocellular carcinoma. However, in case of hepatocellular carcinoma, it is possible for subjects to be enrolled into the study only if the treatment for local lesion was carried out ≥6 months ago and the treated area showed disease progression, or a curatively resectable new lesion has occurred outside the previously treated area, and other inclusion/exclusion criteria are met.
3. Patients with history of other cancers within three years prior to the study treatment. However, patients with other cancers with less influence on their prognosis such as carcinoma in situ or thyroid papillary carcinoma, in the opinion of the investigator, can be enrolled into the study.
4. History of hepatic encephalopathy.
5. Clinically significant ascites defined as follows:

   A. When screening, the physical examination reveals ascites or

   B. Previous ascites that required treatment and continuous prevention or current ascites that require treatment.

   <Investigational medicinal product-related exclusion criteria>
6. History of active autoimmune disease with systematic treatment (i.e. immunomodulator, corticosteroid, or immunosuppressant) required within the past 2 years. Replacement therapy (e.g. physiological corticosteroid replacement therapy due to dysfunction of thyroxine, insulin, adrenal gland, or pituitary gland, etc.) is not regarded as a form of systematic treatment and would be allowed.
7. Diagnosis of immunodeficiency or within 7 days prior to the first administration of investigational medicinal product treatments with chronic systematic steroids (the dose equivalent to 10 mg/day of prednisone) or immunosuppressive therapy in any other forms are not permitted.
8. History of non-infectious interstitial pneumonia requiring treatment of steroids or currently diagnosed.
9. Any prior treatment with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody or other antibodies or drugs, specifically target co-stimulatory T cells or immune checkpoint pathways.

   <General exclusion criteria>
10. Any known hypersensitivity or anaphylaxis of severeness to recombinant proteins containing monoclonal antibodies.
11. Active infection with systematic treatment required.
12. From the viewpoint of the investigator, medical conditions, treatments, or laboratory test abnormalities that are likely to cause confusion in clinical trial results, or that are likely to interfere with subjects' participation throughout the entire study, or that are not considered to be in the best interests of the subjects.
13. Positive urine test or blood pregnancy test in childbearing females within 7 days prior to the first administration of investigational medicinal product.
14. Pregnant or lactating, or during the scheduled study period of 90 days after the final administration of investigational medicinal product, subjects have a plan to have conception.
15. Diagnosis of symptomatic congestive heart failure (i.e. New York Heart Association Classification class II and up) or history of clinically significant heart arrhythmia that requires other antiarrhythmic drugs other than beta blockers and digoxin, or currently diagnosed or occurrence of conduction disorders (atrial fibrillation, paroxysmal supraventricular tachycardia are exceptional) within 6 months prior to the study, active coronary artery diseases, unstable angina, new occurrence of angina within 3 months before enrollment of the study, cardiac infarction within 6 months before enrollment of the study.
16. History of human immunodeficiency virus (HIV 1/2 antibody)
17. Subjects with active hepatitis B (HBsAg-positive or detectable HBV DNA) or hepatitis C (detectable HCV RNA). Patients with hepatitis B can be enrolled in the study, only if HBV DNA <500 IU/mL (or 2500 copies/mL). Patients with positive-HCV antibody can be enrolled only if negative HCV RNA.
18. History of allogeneic tissue/solid organ transplant.
19. Inoculation with live vaccine 28 days prior to the first administration of investigational medicinal product.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2019-09-09 (Actual); Primary Completion 2026-09-09 (Estimated); Study Completion 2026-09-26 (Estimated)

PRIMARY OUTCOMES:
Major pathologic response rate | After surgical resection within 28days
  Evaluation of major pathologic response rate (a proportion of residual viable tumor cells <10%) after administration of pre-operative immune checkpoint inhibitor IMC-001

SECONDARY OUTCOMES:
The safety and feasibility | Within 14 days after the end of Cycle 2 (+,- 4days)
  Evaluation of safety assessed by NCI CTCAE v. 4.03 and evaluation of feasibility assessed by the occurrence of delays in prearranged surgery.
R0 resection rate | After surgical resection within 1 month
  Evaluation of R0 resection rate
Clinical tumor response rate | 1 month
  Evaluation of clinical tumor response rate by RECIST v1.1
Clnical disease control rate | 1 month
  Evaluation of clinical disease control rate by RECIST v1.1
Progression-free survival | 2 years
  Evaluation of progression-free survival
Relapse-free survival | 2 years
  Evaluation of relapse-free survival
Overall survival | 2 years
  Evaluation of overall survival
The rates and patterns of cancer progression/relapse | 2 years
  Evaluation of the rates of cancer progression/relapse
Patterns of cancer progression/relapse | 2 years
  Evaluation of the pattern of cancer progression/relapse

OTHER OUTCOMES:
Discovery of predictive and/or prognostic biomarkers | 2 years
  Discovery of predictive and/or prognostic biomarkers using pre- and post- treatment tumor tissue, blood (circulating tumor DNA, immune cells, etc.), and stool (microbiome) by performing immune profiling and genome analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea